CLINICAL TRIAL: NCT04408326
Title: Efficacy and Safety of Angiotensin II Use in COVID-19 Patients With Acute Respiratory Distress Syndrome
Brief Title: Efficacy and Safety of Angiotensin II Use in Coronavirus Disease(COVID)-19 Patients With Acute Respiratory Distress Syndrome
Acronym: ACES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Australian and New Zealand Intensive Care Research Centre (Other); Monash University (Other); Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 283005
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: COVID; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Angiotensin II; Receptors, Interleukin-6; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Angiotensin II: Patients with COVID-19 and acute respiratory distress syndrome who received angiotensin II as an add-on vasopressor will be collected
  Interventions: Drug: Angiotensin II
- Anakinra: Patients with COVID-19 and acute respiratory distress syndrome who received Anakinra (interleukin 1 receptor antagonist) will be collected
  Interventions: Drug: Interleukin-1 receptor antagonist
- Angiotensin II control: Patients with COVID-19 and acute respiratory distress syndrome who also received vasopressor support will be matched to angiotensin II group by date of intensive care unit admission, age, history of hypertension, history of angiotensin converting enzyme inhibitor/angiotensin receptor blocker, respiratory support
- Anakinra control: Patients with COVID-19 and acute respiratory distress syndrome will be matched to Anakinra group by matching age and date of intensive unit care admission

INTERVENTIONS:
Drug: Angiotensin II — Exogenous angiotensin II acts on angiotensin II type 1 receptor and raise blood pressure by vasoconstriction, salt and water retention, and stimulation of aldosterone hormone
  Groups: Angiotensin II
Drug: Interleukin-1 receptor antagonist — Interleukin-1 receptor antagonist is an immunomodulating drug aiming to mitigate cytokine storm in COVID-19 patients
  Other Names: Anakinra
  Groups: Anakinra

SUMMARY:
This study aims to find out whether the use of angiotensin II, which is a drug to raise blood pressure has been approved by European Medical Agency in August 2019, as an add-on medication to increase blood pressure in patients with COVID-19, acute severe lung injury, inflammation and severe shock, compared with standard medication. In addition, the investigators will collect the data of Anakinra, another drug which is frequently used in this condition to reduce inflammation.

The investigators will collect clinical data and outcomes from critical care patients. The investigators will analyse for whom these drugs are most beneficial and explore whether there are any patients who don't benefit or have side effects.

DETAILED DESCRIPTION:
COVID-19 is a rapidly evolving pandemic with approximately 5% of all patients requiring admission to the intensive care unit. In critically ill patients infected with COVID-19, ARDS is found in 40%, more than 25% require continuous renal replacement therapy, and more than 10% develop vasodilatory shock. Currently, supportive treatment is the mainstay treatment, with fluid administration and vasopressors for haemodynamic support and lung-protective ventilation in patients with severe respiratory failure. Targeted drugs, antiviral therapies, and vaccines are still currently being developed and studied. To date, there is insufficient evidence to recommend any drug over another.

Angiotensin II is a major product of the renin-angiotensin-aldosterone system (RAAS) system. Initially, renin is secreted by hypotension, activation of sympathetic nervous system, and decreased sodium delivery to distal tubules. Renin then stimulates angiotensinogen to be converted into angiotensin I. Angiotensin I is cleaved to angiotensin II by angiotensin-converting enzyme (ACE). ACE is an endothelium-bound ectoenzyme produced by pulmonary endothelium and endothelium from the systemic circulation.

Angiotensin II has a variety of effects, mainly blood pressure elevation via AT-1 receptors, thereby causing direct vasoconstriction, stimulation of vasopressin release for water reabsorption, and stimulation of aldosterone release from the adrenal glands. Angiotensin II is converted to angiotensin(1-7) by angiotensin-converting enzyme 2 (ACE2_. Angiotensin(1-7) has vasodilatory, anti-inflammatory, and anti-apoptotic properties.

The RAAS system may be over- or under-stimulated during sepsis. Diseases that involve pulmonary vasculature e.g. acute respiratory distress syndrome (ARDS) or endotoxaemia can alter ACE function. Studies have shown that patients with lower Ang II and ACE levels were more likely to die. In addition, AT-1 receptors are downregulated from increased inflammatory cytokines, hence diminished vasopressor response in sepsis patients. In COVID-19 patients with ARDS, four mechanisms are proposed in response to deficient functional ACE. First, inadequate production of angiotensin II leads to decreased AT-1 receptor activation, leading to vasodilatation and hypotension. Second, the accumulation of its substrate, angiotensin I, leads to catabolism of angiotensin I into angiotensin(1-7), which causes further vasodilatation. Third, angiotensin(1-7) activates nitric oxide(NO) synthase, stimulates production of NO, another potent vasodilator. Lastly, dysfunctional ACE impairs ACE-dependent hydrolysis of bradykinin, which is another vasodilatory substance. Furthermore, COVID-19 has been shown to bind to the ACE2 receptor for cell entry and viral replication. Angiotensin II has been shown in vitro to downregulate ACE2 by internalization and degradation in both mouse and human models.

Therefore, exogenous angiotensin II is proposed as a potent vasoconstrictor in COVID-19-associated ARDS with vasodilatory shock. Several studies, including a recent randomised controlled trial, have shown angiotensin II as an effective vasopressor. In the largest trial to date, 321 patients were randomized to Ang II (n=163) or placebo (n=158). Most of the included patients had sepsis (80.7%). Patients were included if they were more than 18 years old with vasodilatory shock, defined as mean arterial pressure (MAP) between 55 and 70 mmHg, requiring norepinephrine equivalent dose ≥ 0.2 mcg/kg/min for at least 6 hours, had received at least 25 mL/kg crystalloids within the last 24 hours, and met either of the following criteria; cardiac index more than 2.3 L/min, central venous oxygen saturation (ScvO2) > 70%, or central venous pressure (CVP) > 8 mmHg. Patients who were randomized to Ang II had a higher proportion of meeting MAP target of ≥ 75 mmHg or a ≥ 10 mmHg increase in MAP at 3 hours compared with placebo (69.9% vs 23.4%; p <0.001). Patients who received angiotensin II also had lower noradrenaline requirement at 3 hours and lower cardiovascular SOFA score at 48 hours. Subsequent post-hoc analyses have shown that patients who received Angiotensin II were more likely to be liberated from renal replacement therapy (RRT) within 7 days (38% Ang II versus 15% placebo; p = 0.007). Those who might benefit from Ang II included patients with acute physiologic and chronic health evaluation (APACHE) II score ≥ 30, those with elevated renin and lower baseline Ang II levels, and severe ARDS patients with partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) ratio < 100. In 2019, the European Medical Agency approved angiotensin II as a vasoconstrictor to raise blood pressure in patients with septic or other distributive shock who remain hypotensive despite adequate volume restitution and application of catecholamines and other available vasopressor therapies.

Noradrenaline is currently recommended by the consensus guideline as the first line vasopressor for COVID-19 patients with vasodilatory shock. There is insufficient evidence to issue a treatment recommendation on the use of angiotensin II in critically ill adults with confirmed COVID-19 infection with ARDS and vasodilatory shock. Therefore, this study aims to compare the efficacy of angiotensin II as an add-on vasopressor with optimised standard of care.

Critically ill patients with COVID-19 infection also often receive Anakinra to modulate the inflammatory response. The investigators would also like to collect the data of patients treated with and without Anakinra.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) admitted to intensive care units overseen by critical care consultants
2. Confirmed COVID-19 infection
3. ARDS defined as per the BERLIN ARDS definition1
4. For angiotensin data only: Vasodilatory shock as diagnosed clinically by the treating physicians and receiving noradrenaline for less than 12 hours from the onset of shock or arrival to hospital

Exclusion Criteria:

1. Pure cardiogenic shock
2. Stage 4 cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed COVID-19 infection and acute respiratory distress syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportions of patients with mean arterial pressure ≥ 65 mmHg or an increase of mean arterial pressure ≥10 mmHg at 3 hours | 3 hours
  Percentage

SECONDARY OUTCOMES:
Noradrenaline dose | 1 hour and 3 hours
  microgram/kg/min
Sequential Organ Failure Assessment (SOFA) score | baseline, 24, and 48 hours
  Changes in score, minimum 0, maximum 24, the higher score showing worse prognosis
RRT-free days | 28 days
  Patients who are alive and do not require renal replacement therapy at 28 days
RRT discontinuation | 7 and 28 days
  Proportions of patients who do not require renal replacement therapy
Serum creatinine | 7 days and 28 days
  micromol/L
PaO2/FiO2 ratio | baseline, 24, and 48 hours
  Changes in value
Mortality | 7 days and 28 days
  Mortality rate
Adverse events | 28 days
  e.g. arrhythmia, thromboembolism, etc.
Change in serum C-reactive protein | 7 days
  Change in serum C-reactive protein
Change in serum ferritin | 7 days
  Change in serum ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, Principal Investigator — Department of Critical Care, Guy's & St Thomas' Hospital
Locations (1):
- Guy's & St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided